CLINICAL TRIAL: NCT04317248
Title: Precision Study on "Cocktail" Therapy to Improve the Efficacy of Hepatitis B-related Hepatocellular Carcinoma
Brief Title: "Cocktail" Therapy for Hepatitis B Related Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuehua Huang (Other)
Collaborators: Sun Yat-sen University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor-Investigator, Yuehua Huang, Laboratory director of hepatology，Deputy director of infection, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019B110233002
Record Dates: First submitted 2019-10-07; First posted 2020-03-23 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; hepatitis B; Dendritic cells vaccine; cell therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MSDCV immune therapy combined with radical surgery therapy (Experimental): Multiple Signals loaded Dendritic Cells Vaccine(MSDCV) immune therapy：one time every 4 weeks during 0 weeks to 20 weeks, about 5*10^7 cells per time, total 6 times; Hepatocellular Carcinoma Radical surgery therapy: one time at a good operation time before the first time of MSDCV immune therapy
  Interventions: Drug: Cyclophosphamide; Biological: Multiple Signals loaded Dendritic Cells Vaccine
- Radical surgery therapy (No Intervention): Hepatocellular Carcinoma Radical surgery therapy: one time at a good operation time
- MSDCV immune therapy combined with TACE therapy (Experimental): Multiple Signals loaded Dendritic Cells Vaccine(MSDCV) immune therapy：one time every 4 weeks during 0 weeks to 20 weeks, about 5*10^7 cells per time, total 6 times; Transcatheter Hepatic Arterial Chemoembolization (TACE) therapy: the first time of TACE therapy must perform before the first time of MSDCV immune therapy， then perform when necessary according to subjects condition
  Interventions: Drug: Cyclophosphamide; Biological: Multiple Signals loaded Dendritic Cells Vaccine
- TACE therapy (No Intervention): Transcatheter Hepatic Arterial Chemoembolization (TACE) therapy: perform when necessary according to Subjects condition
- MSDCV immune therapy combined with targeted agents therapy (Experimental): Multiple Signals loaded Dendritic Cells Vaccine(MSDCV) immune therapy：one time every 4 weeks during 0 weeks to 20 weeks, about 5*10^7 cells per time, total 6 times; Targeted agents therapy: Sorafenib or Lenvatinib. For Sorafenib: 0.4g twice daily; for Lenvatinib: 12mg/8mg per day according to subjects condition
  Interventions: Drug: Cyclophosphamide; Biological: Multiple Signals loaded Dendritic Cells Vaccine
- Targeted agents therapy (No Intervention): Targeted agents therapy: Sorafenib or Lenvatinib. For Sorafenib: 0.4g twice daily; for Lenvatinib: 12mg/8mg per day according to subjects condition

INTERVENTIONS:
Drug: Cyclophosphamide — Intravenous drip，250mg/m^2 per time，two days before each times of MSDCV therapy，total 6 times, in order to improve the immunosuppressive microenvironment of tumor，reduce CD4+CD25+FOXP3+regulatory T cells (Tregs）
  Other Names: Endoxan
  Arms: MSDCV immune therapy combined with TACE therapy; MSDCV immune therapy combined with radical surgery therapy; MSDCV immune therapy combined with targeted agents therapy
Biological: Multiple Signals loaded Dendritic Cells Vaccine — one time every 4 weeks during 0 weeks to 20 weeks, about 5*10^7 cells per time, intravenous driptotal 6 times;
  Other Names: MSDCV
  Arms: MSDCV immune therapy combined with TACE therapy; MSDCV immune therapy combined with radical surgery therapy; MSDCV immune therapy combined with targeted agents therapy

SUMMARY:
The effect of anti-tumor treatment is not satisfying in HBV-related hepatocellular carcinoma (HBV-HCC) for reasons that HBV-HCC carries highly heterogeneous antigens to facilitate cancer cells escaping from immune surveillance and constructs an immunosuppressive microenvironment. Correspondingly, multiple signals loaded dendritic cells vaccine can efficiently present T cells with antigens of HCC sensitize their antitumor properties meanwhile low dose cyclophosphamide (CY) can effectively improve the microenvironment of immunity. Therefore, we put forward a new scientific therapy called "multiple signals loaded dendritic cells vaccine combined low dose of cyclophosphamide" combining with radical surgery or TACE or targeted agents for patients with hepatocellular carcinoma to prolong their survival time.

DETAILED DESCRIPTION:
Detailed Description Patients who have good compliance complying with the inclusion criteria will be enrolled into our research. The 600 patients will be randomly assigned to experimental group and control group with the ratio of 1:1, control group will receive radical surgery or TACE or targeted agent treatment solely; another group (experimental group) after enrollment will radical surgery or TACE or targeted agent treatment in the first course. Then 20ml blood is taken for multiple signals loaded dendritic cells (MSDCV) culture (cell culture takes 7 days). Low dose (250mg/m^2) CY treatment will be performed on patients two days before the MSDCV treatment. The MSDCV combined CY therapy will perform per 4 weeks, total 6 times. All patients are evaluated the safety and efficacy of treatment by monitoring their blood parameters, tumor indicators and imaging examinations at each visit.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with AASLD guidelines for the diagnosis of hepatocellular carcinoma，histology or imaging confirmed as primary hepatocellular carcinoma
* Patients with history of hepatitis B infection
* Male and female adult subjects (18～70 years old)
* Patients haven't received radiation therapy or chemotherapy or immunotherapy
* Normal renal function
* Blood routine test: Hb>=9g/dL, white cell count>=1.5*10^9/L, platelet count>=50*10^9/L
* Liver function: bilirubin<=50umol/L, aspartate aminotransferase (AST) or alanine aminotransferase(ALT)<=5 times the upper limit of normal
* Child-Pugh score<=9
* Human Chorionic Gonadotropin(HCG) test negative(-) if patients are women of reproductive ages
* Women of reproductive ages promise to contracept until therapy course has been finished for 3 months
* Patients who have signed up informed consents

Exclusion Criteria:

* Extrahepatic metastasis of hepatocellular carcinoma oHistory of embolism, chemotherapy or radiation
* History of major surgery in last 4 weeks
* History of radiofrequency ablation in last 6 weeks
* Acute infections in last 2 weeks
* Child-Pugh scores>9
* Patients with hepatic encephalopathy
* Patients with ascites needed drainage
* Patients have history of other cancer
* Patients have history of HIV
* Pregnant women
* Patients with severe diseases like cardiac dysfunction
* Patients with mental illness that influence signing informed consents
* HBV infection combined with other types of hepatitis
* Patients with autoimmune diseases
* Immunosuppressant drugs users
* Patients cannot follow our trial principle

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS), month | 240 weeks
  The time from randomization until first documented progression or death from any cause，whichever came first

SECONDARY OUTCOMES:
serum AFP(alpha fetoprotein）, ng/ml | 240 weeks
  Measured for each subjects at each visits
serum PIVKA-II(Protein Induced by Vitamin K Absence or Antagonist-II), μg/L | 240 weeks
  Measured for each subjects at each visits
Overall Survival (OS), month | 240 weeks
  The time from random assignment to death from any cause
tumor size, mm | 240 weeks
  Utilizing Liver CT or MR examination
Number of participants with treatment-related adverse events | 240 weeks
  Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yuehua Huang, doctorate, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (4):
- China (4):
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer center, Guangzhou, Guangdong
  - Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Zhongshan University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No